CLINICAL TRIAL: NCT06308198
Title: A Phase 3, Multicenter, Randomized, Placebo-Controlled Study of AGN-151586 for the Treatment of Moderate to Severe Glabellar Lines
Brief Title: A Study to Evaluate AGN-151586 Intramuscular Injections in Adult Participants for Treatment of Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: M24-008
Record Dates: First submitted 2024-03-07; First posted 2024-03-13 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Glabellar Lines
Keywords: Glabellar Lines; AGN-151586

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Double-Blind Period: AGN-151586 (Experimental): Participants will receive AGN-151586 in the glabellar complex on Day 1.
  Interventions: Drug: AGN-151586
- Double-Blind Period: Placebo (Placebo Comparator): Participants will receive Placebo in the glabellar complex on Day 1.
  Interventions: Drug: Placebo
- Open-Label: AGN-151586 (Experimental): Participants who meet all retreatment criteria will receive AGN-151586 in the glabellar complex on Day 43.
  Interventions: Drug: AGN-151586

INTERVENTIONS:
Drug: AGN-151586 — Intramuscular Injections
  Arms: Double-Blind Period: AGN-151586; Open-Label: AGN-151586
Drug: Placebo — Intramuscular Injections
  Arms: Double-Blind Period: Placebo

SUMMARY:
Facial lines that develop from repeated facial expression, such as glabellar lines (GL), are typically treated by selectively weakening specific muscles with small quantities of botulinum toxin. The purpose of this study is to evaluate the safety and efficacy of AGN-151586 compared to placebo in adult participants.

AGN-151586 is an investigational product being developed for the treatment of GL. In the first period, participants are randomly assigned to receive AGN-151586 or placebo. Each group receives a different treatment. There is a 1 in 3 chance that participants will be assigned to placebo. In the second period, all participants who meet retreatment criteria will receive open-label AGN-151586. Around 160 participants will be enrolled in the study at approximately 14 sites in China, Taiwan, and Japan.

Participants will receive either AGN-151586 or Placebo administered as 5 intramuscular injections to the glabellar complex on Day 1. Eligible participants may then receive AGN-151586 injections on Day 43 and will be followed for up to 6 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care due to multiple study visits. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must have Moderate or severe glabellar lines (GL) at maximum frown as assessed by both the investigator and participant using the FWS-A at Screening and Baseline Day 1 visit. The investigator and participant ratings must match within a visit but do not have to match between Screening and Baseline Day 1.
* Must be in good health as per investigator's judgment based on medical history, physical examination, and vital sign measurements.

Exclusion Criteria:

* Uncontrolled systemic disease.
* Infection or dermatological condition at the treatment injection sites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-02-26 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a >= 2-Grade Improvement from Baseline on the Facial Wrinkle Scale with Asian (FWS-A) Guide According to Investigator Assessment of Glabellar Lines (GL) Severity at Maximum Frown | Day 7
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants with a >= 2-Grade Improvement from Baseline on the FWS-A Guide According to Participant Assessment of GL Severity at Maximum Frown | Day 7
  Participants' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Number of Participants with Adverse Events (AEs) | Up to approximately Day 84
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants with a >= 2-Grade Improvement from Baseline on the FWS-A Guide According to Participant Assessment of GL Severity at Maximum Frown | Hour 24
  Participant's assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants with a >= 2-Grade Improvement from Baseline on the FWS-A Guide According to Investigator Assessment of GL Severity at Maximum Frown | Hour 24
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants Achieving Mostly satisfied or Very satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Follow-Up Version Item 5 (overall satisfaction) for GL | Hour 24
  The FLSQ consists of 13 questions that assess treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with GL using the FLSQ 5-point scale ranging from Very dissatisfied to Very satisfied. Follow-up Item 5 (satisfaction with the effect of treatment) can also be used as a stand-alone item.
Percentage of Participants Achieving Mostly satisfied or Very satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Follow-Up Version Item 4 (natural look) for GL | Day 7
  The FLSQ consists of 13 questions that assess treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with GL using the FLSQ 5-point scale ranging from Very dissatisfied to Very satisfied. Follow-up Item 4 (satisfaction with the natural look) can also be used as a stand-alone item.
Percentage of Participants Achieving Mostly satisfied or Very satisfied on the Facial Line Satisfaction Questionnaire (FLSQ) Follow-Up Version Item 5 (overall satisfaction) for GL Over Time | Baseline up to approximately Day 84
  The FLSQ consists of 13 questions that assess treatment satisfaction and psychosocial impact. Participants assessed their satisfaction with GL using the FLSQ 5-point scale ranging from Very dissatisfied to Very satisfied. Follow-up Item 5 (satisfaction with the effect of treatment) can also be used as a stand-alone item.
Double-Blind Period: Time to the First >= 1-Grade Improvement from Baseline on the FWS-A According to Participant Assessment of GL Severity at Maximum Frown | Baseline to Day 42
  Participants' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Double-Blind Period: Time to the First >= 1-Grade Improvement from Baseline on the FWS-A According to Investigator Assessment of GL Severity at Maximum Frown | Baseline to Day 42
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Double-Blind Period: Percentage of Participants with a >= 2-Grade Improvement from Baseline on the FWS-A Guide According to Participant Assessment of GL Severity at Maximum Frown Over Time | Baseline to Day 42
  Participants' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Double-Blind Period: Percentage of Participants with a >= 2-Grade Improvement from Baseline on the FWS-A Guide According to Investigator Assessment of GL Severity at Maximum Frown Over Time | Baseline to Day 42
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Double-Blind Period: Time to Loss of None or Mild FWS-A According to Participant Assessment of FWS-A at Maximum Frown | Baseline to Day 42
  Participants' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Double-Blind Period: Time to Loss of None or Mild FWS-A According to Investigator Assessment of FWS-A at Maximum Frown | Baseline to Day 42
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants Achieving None or Mild on the FWS-A According to Participant Assessment Using FWS-A at Maximum Frown Over Time | Baseline to Day 84
  Participants' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants Achieving None or Mild on the FWS-A According to Investigator Assessment Using FWS-A at Maximum Frown Over Time | Baseline to Day 84
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants with a >= 1-Grade Improvement from Baseline on FWS-A According to Participant Assessment of GL Severity at Maximum Frown | Hour 24
  Participants' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants with a >= 1-Grade Improvement from Baseline on FWS-A According to Investigator Assessment of GL Severity at Maximum Frown | Hour 24
  Investigators' assessments of the severity of GL using the 4-grade FWS-A, where 0=none and 3=severe. Higher grades indicate more severity.
Percentage of Participants with a >= 20-Point Improvement from Baseline in 11-Item Facial Line Outcomes (FLO-11) Total Scores (transformed) for GL | Day 7
  The FLO-11 Questionnaire consists of 11 questions that assess appearance-related psychological impact. Participants assessed their satisfaction with GL using the FLO-11 11-item scale that ranges from 0 (Not at all) to 10 (Very much) with higher scores indicating negative impact. Total scores are transformed to a 0 to 100 scale, with higher scores indicating better psychosocial outcomes.
Percentage of Participants with a >= 4-Point Improvement from Baseline in 11-Item FLO-11 Item 10 (look angry) for GL | Day 7
  The FLO-11 Questionnaire consists of 11 questions that assess appearance-related psychological impact. Participants assessed their satisfaction with GL using the FLO-11 11-item scale that ranges from 0 (Not at all) to 10 (Very much) with higher scores indicating negative impact.
Percentage of Participants with a >= 4-Point Improvement from Baseline in 11-Item FLO-11 Item 5 (look less attractive) for GL | Day 7
  The FLO-11 Questionnaire consists of 11 questions that assess appearance-related psychological impact. Participants assessed their satisfaction with GL using the FLO-11 11-item scale that ranges from 0 (Not at all) to 10 (Very much) with higher scores indicating negative impact.
Percentage of Partcipatns who Achieve Patient-Reported Global Assessment of Change in GL Based on the Global Assessment of Change in Glabellar Lines (GAC-GL) Over Time | Baseline up to approximately Day 84
  The GAC-GL Questionnaire is a 2-item measure that assesses the appearance of the participant's GL "now" in comparison with their perspective before treatment at rest and at maximum furrow. The response options are scored on a 7-point VDS ranging from Very much improved to Very much worse. Scores are unique for at rest and maximum contraction, and they are simply the responses to the items.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (12):
- China (9):
  - Beijing Hospital /ID# 256084, Beijing, Beijing Municipality
  - Dermatology Hospital of Southern Medical University /ID# 256172, Guangzhou, Guangdong
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 255871, Wuhan, Hubei
  - Nanjing Drum Tower Hospital /ID# 255936, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University /ID# 255937, Nanjing, Jiangsu
  - Wuxi People's Hospital /ID# 256029, Wuxi, Jiangsu
  - Xianyang Hospital of Yan'an University /ID# 256774, Xianyang, Shaanxi
  - Huashan Hospital, Fudan University /ID# 255870, Shanghai, Shanghai Municipality
  - Zhejiang Provincial People's Hospital /ID# 256028, Hangzhou, Zhejiang
- Tokyo Center Clinic /ID# 267380, Chuo-ku, Tokyo, Japan
- Taiwan (2):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 260669, Kaohsiung City
  - Tri-Service General Hospital /ID# 260673, Taipei

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-008